CLINICAL TRIAL: NCT05448560
Title: BRidging Information Divides and Gaps to Ensure Survivorship: the BRIDGES Randomized Controlled Trial of a Multilevel Intervention to Improve Adherence to Childhood Cancer Survivorship
Brief Title: A Multilevel Intervention to Improve Adherence to Childhood Cancer Survivorship
Acronym: BRIDGES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Colorado, Denver (Other); Hackensack Meridian Health (Other); NYU Langone Health (Other); Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01CA261881 (NIH)
Record Dates: First submitted 2022-06-16; First posted 2022-07-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Childhood Cancer; Survivorship; Health Care Utilization; Health Knowledge, Attitudes, Practice; Adherence, Patient
Keywords: childhood cancer survivors; survivorship care; randomized controlled trial
MeSH Terms: conditions — Neoplasms; Patient Acceptance of Health Care; Behavior; Patient Compliance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-level Intervention of shared model of survivorship care (Experimental): 1. Patient survivorship education via telehealth with the cancer center
  2. Ongoing patient-tailored education program by MyChart within the EHR patient portal
  3. Structured interactive phone communication between the research RN at the cancer center and community PCP clinic
  4. In-person visit with the PCP clinic for survivorship care.
  Interventions: Behavioral: Multi-level Intervention of shared model of survivorship care
- "Gold standard" cancer center-based survivorship clinic (Active Comparator): In-person visit at specialty survivorship clinic
  Interventions: Other: Comparison Group

INTERVENTIONS:
Behavioral: Multi-level Intervention of shared model of survivorship care — 1) Patient survivorship education via telehealth with the cancer center- The research registered nurse (RN) will discuss the contents of the survivorship care plan and coordination between the cancer center and PCP clinic. 2) Ongoing patient-tailored education program by MyChart within the EHR patient portal- Patients will be asked to select survivorship topics of interest from a panel (e.g. school issues, fertility, fatigue, physical activity, single kidney health, emotions/coping) that will then be sent over 1 year. 3) Structured interactive phone communication between the research RN at the cancer center and community PCP clinic- The discussion will explain the patient's cancer history, tumor recurrence monitoring schedule, individualized risk of late effects and surveillance schedule, psychosocial challenges, health behaviors, and coordination between the cancer center and PCP clinic. 4) In-person visit with the PCP clinic for survivorship care.
  Arms: Multi-level Intervention of shared model of survivorship care
Other: Comparison Group — Participants will be contacted by study staff at their cancer center to schedule an in-person visit at the survivorship clinic that will include a comprehensive history focused on cancer-related medical and psychosocial issues, physical examination, ordering of recommended surveillance for late effects, and delivery of hard copy of their survivorship care plan.
  Arms: "Gold standard" cancer center-based survivorship clinic

SUMMARY:
More than 80% of childhood cancer survivors develop serious or life-threatening late effects after cancer therapy, but <20% receive recommended survivorship care offered at cancer center survivorship clinics. In a shared care model, the investigators propose to investigate an innovative multi-level intervention consisting of: 1) patient survivorship education via telehealth with the cancer center, 2) ongoing patient-tailored education program within the electronic health record patient portal, 3) a structured interactive phone communication between the cancer center and the primary care clinic, and 4) an in-person visit with the primary care clinic for survivorship care with the goal of achieving high rates of adherence to recommended surveillance for late effects, as well as improving patient and physician knowledge and self-efficacy. If this scalable intervention demonstrates patient completion of recommended care comparable to cancer center survivorship clinics, this innovative study has the enormous potential to deliver recommended care to a larger proportion of childhood cancer survivors and reduce survivorship care disparities, while engaging p to integrate survivorship care as part of overall, lifelong health maintenance.

DETAILED DESCRIPTION:
More than 80% of childhood cancer survivors (CCS) develop serious or life-threatening late effects. Yet <20% of CCS receive recommended survivorship care, despite the availability of consensus guidelines for lifelong surveillance for late effects starting 2 years post-therapy. The "gold standard" cancer center-based survivorship clinic provides high-quality care to CCS who attend, but patients avoid reminders of their past cancer and lack knowledge and self-efficacy for survivorship care. Other barriers include travel distance, inadequate insurance, and out-of-pocket costs-these structural issues contribute to health disparities. Partnering with community primary care provider (PCP) clinics in a shared model of care is a promising strategy to overcome these barriers, but PCPs lack knowledge, self-efficacy, and interactive communication with the cancer center and are confused about the division of care responsibilities. This intervention is scalable and distance-based, is informed directly by patient and PCP barriers and preferences from previous studies, and is boosted by a nationwide explosion in telehealth services precipitated by the COVID-19 crisis. The proposed randomized controlled trial will enroll 240 CCS 2.0-4.0 years post-chemotherapy/radiation to investigate an innovative multi-level intervention (i.e., interpersonal and organizational levels) consisting of 1) patient survivorship education via telehealth with the cancer center, 2) ongoing patient-tailored education program within the electronic health record (EHR)'s patient portal, 3) a structured interactive phone communication between the cancer center and the PCP clinic (with 1-year follow-up call), and 4) an in-person visit with the PCP clinic for survivorship care. The comparison group will be randomized to an in-person visit with their cancer center survivorship clinic. This study includes 4 centers with high proportions of subgroups vulnerable to survivorship care disparities (i.e., rural, Black, Latinx, Spanish-speaking, socioeconomically disadvantaged). Both groups will be asked to begin recommended surveillance for late effects within 1-year post-randomization, separate from tumor recurrence monitoring by the primary oncologist. The Specific Aims are to Aim 1- Demonstrate patient completion of guideline-recommended surveillance tests in intervention participants is not inferior, i.e. within 10%, to that in the comparison group; Aim 2- Achieve greater 1) patient knowledge, self-efficacy, and activation and 2) PCP knowledge and self-efficacy with survivorship care among intervention participants and their PCPs compared to the comparison group; and Aim 3- Ascertain process outcomes for the 1) patient and 2) PCP clinic. Outcomes will also be assessed among subgroups with survivorship care disparities. Transformative Impact: If the intervention demonstrates patient completion of recommended survivorship care comparable to cancer center survivorship clinic, the study has the enormous potential to deliver recommended lifelong care to a larger proportion of CCS and reduce survivorship care ies, while engaging patients and PCPs to integrate survivorship care as part of overall, lifelong health maintenance.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with any cancer at age <21 years
2. Treated with chemotherapy and/or radiation
3. 2.0-4.0 years status post-completion of all cancer-related therapy
4. Cancer-free with a life expectancy of ≥2 years
5. English- or Spanish-speaking (also applies to parent/guardian if patient age <18 years)
6. No previous attendance at a specialty survivorship clinic
7. Followed at one of the 4 participating sites: Hackensack, University of North Carolina- Chapel Hill (UNC), University of Colorado Denver (CU), Miller's Children's and Women's Hospital Long Beach (MCWH)

Exclusion Criteria:

* Active medical problems severe enough to not be eligible for receiving survivorship care with primary care provider at the time of recruitment

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient completion of guideline-recommended surveillance tests for late effects of therapy | 1-year post-randomization
  The investigators will assess adherence to surveillance recommended by the Children's Oncology Group Long-term Follow-up Guidelines. The primary analysis will be on tests completed by patients, and not just ordered by physicians, because that is the most meaningful indicator of patient adherence to guidelines
Patient completion of guideline-recommended surveillance tests for late effects of therapy | 2 years post-randomization
  The investigators will assess adherence to surveillance recommended by the Children's Oncology Group Long-term Follow-up Guidelines. The primary analysis will be on tests completed by patients, and not just ordered by physicians, because that is the most meaningful indicator of patient adherence to guidelines

SECONDARY OUTCOMES:
Patient Knowledge: | 1-year post-randomization
  Patient Knowledge Survey developed by Kadan-Lottick et al. for the Childhood Cancer Survey Study which is a 9-item survey regarding treatment history, risk of late effects, need for survivorship care, and purpose of the survivorship care plan. Note that results will not be reported on a scale.
Patient Knowledge: | 2-years post-randomization
  Patient Knowledge Survey developed by Kadan-Lottick et al. for the Childhood Cancer Survey Study which is a 9-item survey regarding treatment history, risk of late effects, need for survivorship care, and purpose of the survivorship care plan. Note that results are not reported on a scale.
Patient Healthcare Self-Efficacy | 1-year post-randomization
  Stanford Chronic Disease Self-Efficacy Scale (score range 1-10, higher score indicates greater self-efficacy) to be administered to patients and proxies
Patient Healthcare Self-Efficacy | 2-years post-randomization
  Stanford Chronic Disease Self-Efficacy Scale (score range 1-10, higher score indicates greater self-efficacy) to be administered to patients and proxies
Patient Activation | 1-year post-randomization
  The 13-item Patient Activation Measure (PAM) will be administered to participants to evaluate the level of patient activation, i.e. patient self-reported knowledge, skill, and confidence for self-management of one's health or chronic condition. Scores range from 0-100 with higher scores reflecting greater patient activation.
Patient Activation | 2-years post-randomization
  The 13-item Patient Activation Measure (PAM) will be administered to participants to evaluate the level of patient activation, i.e. patient self-reported knowledge, skill, and confidence for self-management of one's health or chronic condition. Scores range from 0-100 with higher scores reflecting greater patient activation.
PCP Knowledge and Self-Efficacy | 1-year post-randomization
  Survey consisting of questions regarding the PCPs' familiarity with the surveillance guidelines and confidence in providing survivorship care. Note that results are not reported on a scale.
PCP Knowledge and Self-Efficacy | 2-years post-randomization
  Survey consisting of questions regarding the PCPs' familiarity with the surveillance guidelines and confidence in providing survivorship care. Note that results are not reported on a scale.
Process Outcomes for Patients | 1-year post-randomization
  Patients will complete a survey regarding process outcomes (i.e., feasibility, fidelity, acceptability) associated with the multi-level intervention. Note that results are not reported on a scale.
Process Outcomes for Primary Care Physicians | 1-year post-randomization
  Primary care physicians will complete a survey regarding process outcomes (i.e., feasibility, fidelity, acceptability) associated with the multi-level intervention. Note that results are not reported on a scale.

OTHER OUTCOMES:
Post-intervention qualitative interviews of participants and PCPs | 1-year post-randomization
  The investigators will conduct semi-structured, qualitative interviews with 1) 40 intervention participants and 2) 40 PCP clinics to generate feedback regarding the intervention (e.g. timing, duration, usability). Interviews will explore acceptability of the intervention and how to improve intervention efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kadan-Lottick, MD, MSPH, Principal Investigator — Georgetown Lombardi Comprehensive Cancer Center
Locations (4):
- United States (4):
  - MemorialCare Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Colorado, Denver, Colorado
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of North Carolina Children's Hospital, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
The proposed research will include data from 240 survivors of childhood cancer. The dataset will include (1) demographic data; (2) cancer diagnosis and treatment data; (3) adherence to survivorship care data; (4) knowledge, self-efficacy, and activation data; and (5) process outcomes (feasibility, fidelity, acceptability) data. In compliance with the National Institutes of Health Principles and Guidelines document, the investigators will readily provide all relevant protocols, publications, and the underlying primary data (to the extent possible as guided by the IRB) supporting publications to other academic investigators upon request. To maintain the privacy of the human subjects, data will de-identified. Should any intellectual property arise that requires a patent, the investigators will ensure that the technology (materials and data) remains widely available to the academic research community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After analysis and publication of data addressed in the the aims set forth in R01 CA261881
Access Criteria: Request to study investigators and compliance with all IRB and institutional data usage agreement requirements.

REFERENCES:
- [Derived] Ross WL, Santiago-Rivera Y, Tan MT, Roy MM, Bryant S, Appel BE, Casillas J, Demedis J, Smitherman AB, Horwitz LI, Hurtado-de-Mendoza A, Mendoza JA, Santacroce SJ, Kadan-Lottick NS. Design and methods of a multi-level intervention to improve adherence to childhood cancer survivorship care by partnering with primary care providers: The BRIDGES randomized controlled trial. Contemp Clin Trials. 2025 May;152:107859. doi: 10.1016/j.cct.2025.107859. Epub 2025 Feb 21. PMID 39987960
- See also: NIH Reporter listing of this funded study by the National Cancer Institute — https://reporter.nih.gov/search/6GbyUJneWUuTdw9vdewrUA/project-details/10274932